CLINICAL TRIAL: NCT05157529
Title: AQUABEAM® Robotic System and Ultrasound Accessories (AQUA Study)
Brief Title: AQUABEAM® Robotic System and Ultrasound Accessories
Acronym: AQUA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: PROCEPT BioRobotics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-10283
Record Dates: First submitted 2021-11-19; First posted 2021-12-15 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Benign Prostatic Hyperplasia; Lower Urinary Tract Symptoms
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Intervention Model Description: Prospective single-arm investigational clinical trial assessing the efficacy and safety of the new generation of the AQUABEAM Robotic System (P1G3) and the Apogee 2300 Ultrasound System.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Aquablation (Experimental): The participant will undergo aquablation procedure for Benign Prostate Hypeplasia (BPH) treatment using the AQUABEAM Robotic System and Ultrasound Accessories
  Interventions: Device: AQUABEAM Robotic System; Device: Apogee 2300 digital color doppler ultrasound imaging system

INTERVENTIONS:
Device: AQUABEAM Robotic System — The AQUABEAM Robotic System is developed and manufactured by PROCEPT BioRobotics, Corp. It is intended for use in patients suffering from lower urinary tract (LUTS) resulting from benign prostatic hyperplasia (BPH). The AQUABEAM Robotic System is designed for cutting of prostate tissue during minimally invasive surgical procedure and shall be inserted via transurethral approach and is advanced through the urethra and into the prostatic urethra.
  The system is designed to utilize a high-velocity sterile saline stream as the cutting medium which is projected through a nozzle positioned within the prostatic urethra. The nozzle assembly motion is driven by a motor system, controlled by the user. The pressure is generated by a high-velocity pump system controlled by the AQUABEAM Console. The user is allowed to adjust the desired flow rates manually. All functions are displayed on a medical panel computer. Pre-condition parameters are set on the console before operation.
Device: Apogee 2300 digital color doppler ultrasound imaging system — The SIUI Apogee 2300 is a digital ultrasound imaging system capable of the following operating modes: B-Mode (B, 2B, 4B), M-Mode, CFM, CPA, PWD, CWD, Combined (B, M, CFM, CPA, PWD, CWD, XBeam, Panoscope), others (3D, 4D, Trapezoidal /Extended Sector Imaging, Elastography, Anatomical M-mode, TDI, MFI, ECG, VS Flow, Color M, DICOM).
  The system is designed for use in linear, convex, phased array and 3D scanning modes and supports linear, convex, phased array, 3D and endocavity (trans-vaginal and trans-rectal) transducers. The system has cine review, image zoom, measurements and calculations, image storage and review, printing and recording capabilities.

SUMMARY:
Lower urinary symptoms (LUTS) affect many older men and their frequency and severity increase with age. In the age group between 65 and 79 years the rate of men with moderate and severe LUTS is 20 - 25% (Hunter et al. 1994). The complaints are potentially associated with a considerable impairment of the quality of life (Trueman et al. 1999). LUTS in older men are commonly caused by a bladder outlet obstruction (BOO) secondary to benign prostatic enlargement (BPE). The histological term "benign prostatic hyperplasia" (BPH) is frequently used in literature and clinical practice as a synonym for this diagnosis.

Surgical therapy of BPH has continuously evolved in recent years. One of the latest technologies for transurethral prostate desobstruction is the Aquablation therapy, first described in 2015 (AQUABEAM®, PROCEPT BioRobotics, Redwood Shores, CA, USA) (Faber et al 2015). The AQUABEAM Robotic System is the first and only image-guided, heat-free robotic therapy for the treatment of lower urinary tract symptoms (LUTS) due to benign prostatic hyperplasia (BPH). It is designed for cutting of prostate tissue during a minimally invasive surgical procedure. Once inserted via a transurethral approach and advanced through the urethra and into the prostatic urethra, the device applies an ultrasound-guided water jet that precisely ablates the prostate tissue. Aquablation therapy is unique in that it combines cystoscopic visualization, ultrasound imaging and advanced planning software to provide the surgeon with a multidimensional view of the treatment area. This enables personalized treatment planning for the patient's unique anatomy, improved decisionmaking and real-time monitoring during the procedure.

This prospective single-arm investigational clinical trial aims at assessing the efficacy and safety of the new generation of the AQUABEAM Robotic System (P1G3) and the Apogee 2300 Ultrasound System and compare the percentage of patients who are discharged the day of the surgery among different groups of BPH patients who undergo aquablation using the third generation of the AQUABEAM Robotic System.

DETAILED DESCRIPTION:
A- Background:

Lower urinary symptoms (LUTS) affect many older men and their frequency and severity increase with age. In the age group between 65 and 79 years the rate of men with moderate and severe LUTS is 20 - 25%. This rate increases to 90% in men over 80 years old. The complaints are potentially associated with a considerable impairment of the quality of life. LUTS in older men are commonly caused by a bladder outlet obstruction (BOO) secondary to benign prostatic enlargement (BPE). The histological term "benign prostatic hyperplasia" (BPH) is frequently used in literature and clinical practice as a synonym for this diagnosis.

Surgical therapy of BPH has continuously evolved in recent years. Transurethral resection of the prostate (TUR-P) is the current gold standard for the endoscopic management of small to medium prostate volumes. The development of laser-assisted transurethral and other innovative techniques (e.g. REZUM, UROLIFT) have supplemented the surgical spectrum. For large prostate volumes above 80 mL, transurethral laser enucleation (holmium, thulium) is widely established in clinics as an alternative to conventional open surgical simple prostatectomy.

One of the latest technologies for transurethral prostate desobstruction is the Aquablation therapy, first described in 2015 (AQUABEAM®, PROCEPT BioRobotics, Redwood Shores, CA, USA). The device applies an ultrasound-guided water jet that precisely ablates the prostate tissue. The second generation of this robot-assisted system is CE-certified and gained market access in Australia, New Zealand, Canada, and the United States. This device for this study is the third generation of the AQUABEAM Robotic System, which is currently only commercialized in the US.

In recent years, the technology has been evaluated in a total of three monocentric and three multicentric prospective studies. So far, one randomized controlled trial (RCT) has been conducted - the WATER study. The multi-center study, designed as a double-blind, randomized controlled trial, compares the Aquablation therapy with the gold standard TUR-P in small and medium prostate sizes (30-80 mL). The primary endpoint was defined as IPSS change 6 months postoperatively. The primary safety endpoint was stated as the rate of adverse events three months after surgery with a Clavien-Dindo grade ≥ 2 or a Clavien-Dindo grade 1 with persistent dysfunctions such as incontinence, erectile dysfunction or ejaculation disorders. The WATER study confirmed the non-inferiority of the Aquablation therapy regarding the two primary endpoints. The results for the secondary endpoints erectile function (IIEF) and ejaculatory function (MSHQ-EjD) were significantly better in the Aquablation-arm. Interestingly, a subgroup analysis of the WATER patient collective revealed significantly better results regarding IPSS reduction, the primary safety endpoint and the rate of postoperative anejaculation for patients with medium prostate volumes (50-80 mL).

To date, the only prospective study focusing on large prostate volumes is the WATER II trial. In the multi-center and single-arm study design, the safety and efficacy of the procedure was investigated for prostate sizes between 80 and 150 mL. The 1-year follow-up data were published in July 2019. The functional outcome in terms of IPSS reduction, quality of life improvement and Qmax improvement was comparable to previously published data of laser enucleation. The incontinence rate was lower com-pared to the published data for holmium laser enucleation and comparable to the data for open surgical prostate adenoma enucleation. Bleeding complications with necessary blood transfusion were less frequent compared to the data for open surgery but more frequent compared to the data for holmium laser enucleation. In 81% of the sexually active men in this collective, antegrade ejaculation was maintained, which significantly exceeds the published data of the alternative techniques. The main advantage of the method is the short operation time. Since the time of the resection itself is only margin-ally extended as the prostate volume increases, the time advantage is particularly pronounced in the treatment of large prostates. In the WATER II study, the mean procedure time was 37 min (mean resection time: 7.8 min) and was thus significantly shorter than the published data for open surgery (95 min) and laser enucleation (91 min).

The safety and effectiveness of the device has been established in the previous generation of the device: AQUABEAM Robotic System P1G2. The P1G3 system is considered substantially equivalent to the P1G2 system. The indications for use, intended patient population, intended user, safety and efficacy profile of the device remains unchanged for P1G3 compared to P1G2.

B- Clinical experience:

The safety and effectiveness of the AQUABEAM Robotic System P1G3 is equivalent to System P1G2, which has been evaluated in two pivotal US FDA IDE trials, the WATER study (ClinicalTrials.gov ID: NCT02505919), and the WATER II study (ClinicalTrials.gov ID: NCT03123250).

* The WATER study was a prospective multi-center randomized double-blind clinical trial comparing Aquablation of the prostate with the AQUABEAM Robotic System with standard transurethral resection of the prostate (TURP) for the treatment of Lower Urinary Tract Symptoms (LUTS) in prostate size 30-80 cc. One hundred and eighty-four (184) study subjects were randomized at the ratio of 2:1 (Aquablation: TURP). The primary endpoint was defined as IPSS change 6 months postoperatively. The primary safety endpoint was stated as the rate of adverse events three months after surgery with a Clavien-Dindo grade ≥ 2 or a Clavien-Dindo grade 1 with persistent dysfunctions such as incontinence, erectile dysfunction or ejaculation disorders. The WATER study confirmed the non-inferiority of the AQUABEAM Robotic System regarding the two primary endpoints. The results for the secondary endpoints erectile function (IIEF) and ejaculatory function (MSHQ-EjD) were significantly better in the Aquablation-arm. Interestingly, a subgroup analysis of the WATER patient collective revealed significantly better results regarding IPSS reduction, the primary safety endpoint and the rate of postoperative anejaculation for patients with medium prostate volumes (50-80 cc). Three-year study data from the study provided high-quality evidence of the Aquablation therapy for LUTS due to BPH in men with prostate sized between 30 and 80 cc with clinical efficacy and durability similar to TURP.
* To date, the only prospective study focusing on large prostate volumes is the WATER II study. In the multicenter and single-arm study design, the safety and efficacy of the procedure was investigated for prostate sizes between 80 and 150 cc. The 1-year follow-up data were published in July 2019. The functional outcome in terms of IPSS reduction, quality of life improvement and Qmax improvement was comparable to previously published data of laser enucleation. The incontinence rate was lower compared to the published data for holmium laser enucleation and comparable to the data for open surgical prostate adenoma enucleation. Bleeding complications with necessary blood transfusion were less frequent compared to the data for open surgery but more frequent compared to the data for holmium laser enucleation. In 81% of the sexually active men in this collective, antegrade ejaculation was maintained, which significantly exceeds the published data of the alternative techniques. The main advantage of the method is the short operation time. Since the time of the resection itself is only marginally extended as the prostate volume increases, the time advantage is particularly pronounced in the treatment of large prostates. In the WATER II study, the mean procedure time was 37 min (mean resection time: 7.8 min) and was thus significantly shorter than the published data for open surgery (95 min) and laser enucleation (91 min). The Aquablation procedure is a safe and effective, robotically executed and globally reproducible surgical option for the treatment of BPH-related LUTS in men with large prostate glands with continued durable outcomes at 3 years coupled with short operative times, limited hospitalization and low retreatment rates.

C- Clinical investigation design

1. Objectives: Determine the safety and effectiveness of the surgical treatment of lower urinary tract symptoms (LUTS) due to benign prostatic hyperplasia (BPH) when using the AQUABEAM Robotic System P1G3 and Apogee 2300 Ultrasound System.
2. Sample size: Minimum fifty (50) subjects will be enrolled and treated in the study. Up to an additional 10 subjects may be enrolled and treated as roll-in subjects to familiarize the surgeon with the AQUABEAM Robotic System P1G3 prior to treating the study subject.
3. Study duration: Enrollment is expected to take 12 months. Each subject is followed post-operatively through 3 months.

   Note the investigation for the Apogee 2300 ultrasound system and accessories is considered completed after the enrollment goal is achieved and all subjects are discharged.

   Total study duration from the first subject enrolled to the last subject completing the last study follow-up visit is expected to take less than two years.
4. Number of sites: At minimum 1 clinical site in Canada will participate in the study.
5. Point of enrollment: Each patient will be assigned a study ID after signing the informed consent form.

   * Investigators will be responsible for obtaining consent using the current study-specific, REB-approved consent documents prior to any baseline testing for eligibility that goes beyond standard care.
   * Reasons for screen fail will be recorded in study specific form (e.g., did not meet study selection criteria; decline further participating in the study prior to treatment, etc.).
   * Participants will be consented in a manner understandable by the intended patient population and providing adequate time to address any questions or concerns.
   * Documentation of the consenting process and the signed/dated consent documents will be filed in the study Trial Master File.

   An informed consent form must be signed by each patient prior to study enrollment. Informed consent will be obtained according to the Declaration of Helsinki ("Ethical Principles for Medical Research Involving Human Subjects", The World Medical Association Declaration of Helsinki (64th WMA General Assembly, Fortaleza, Brazil, October 2013), requirements of the standard ISO 14155:2020 ("Clinical investigation of medical devices for human subjects-Good clinical practice"), and individual institution guidelines.

   Re-consent will be required where changes are implemented, new information becomes available, or as required by regulations, and re-consent is needed.
6. Study visits and exams:

6.1. Study visits: Screening and Baseline visit: Potential study participants will undergo screening at the study center. Patients must avoid taking non-steroidal anti-inflammatory agents (NSAIDs) or antiplatelet agents (e.g., aspirin, clopidogrel) prior to surgery per standard of care.

Surgical procedure visit: Aquablation therapy will be performed under general or spinal anesthesia at the operating surgeon's discretion. The study surgical procedures will be performed within 90 days of baseline tests.To minimize bleeding, focal cauterization and resection of ablated tissue should be performed for all subjects following the AQUABEAM Handpiece removal. At the end of the procedure, a foley catheter should be placed, continuous bladder irrigation (CBI) should be initiated immediately following the catheter placement and shall continue in the PACU for up to 4 hours. If the degree of hematuria is not clinically significant (grade I-III) after clamping irrigation, subjects will be discharged home. A decision algorithm will be used to discharge subjects. If a patient was discharged home with a catheter, the catheter will be removed at the investigational site.

Follow-up visit: All subjects in this study are intended to be discharged the same day of the Aquablation procedure. The subject will return at 3 months for a final follow up visit, which concludes the subject's participation in the study.

6.2. Study assessments (standard of care): All are considered standard examinations prior to transurethral prostate tissue resection surgery.

Uroflow (Qmax) and PVR: at baseline and the 3-month follow-up visit, the subject will undergo measurement of urinary flow rate (Qmax), urinary mean flow rate (Qmean), total voided volume (TVV), and post-void residual volume (PVR). For a uroflow test to be valid, the voided volume must be ≥ 125 ml. If the total voided volume is less than 150mL, the voided volume must be equal to or greater than 50% of the bladder capacity (defined as voided volume + PVR). The patient can repeat the test if necessary.

International Prostate Symptom Score (IPSS): IPSS is a validated measure of urinary symptoms due to BPH. Subjects will complete an IPSS form at baseline and at the 3-month follow-up visit.

Transrectal ultrasound (TRUS): TRUS is performed to measure patient's prostate size at baseline.TRUS should be performed using the site's standard ultrasound equipment

D- Risk/benefit analysis

Potential benefits: The primary potential benefit of participation is the potential occurrence of successful treatment of lower urinary tract symptoms using the AQUABEAM Robotic System. Additional benefits may be decreased need for urinary catheter postoperatively, faster overall recovery, improved urinary flow and lower residual volumes, low rate of postoperative incontinence and maintenance of ejaculatory function In a patient with urinary retention, the need for catheter use (indwelling or intermittent) may be reduced.

Potential risks: As with any surgical urologic procedure, potential risks of the Aquablation procedure include:

* Anesthesia risk
* Bladder or prostate capsule perforation
* Bladder neck contracture
* Bleeding
* Bruising
* Dysuria
* Electric shock/burn
* Embolism
* Incontinence or overactive bladder
* Infection
* Penile or pelvic pain
* Rectal incontinence / perforation
* Sexual dysfunction, including ejaculatory and erectile dysfunction
* TUR syndrome
* Urethral damage causing false passage or stricture
* Urinary Retention

Risk mitigation: The following steps have or will be taken by the manufacturer and sponsor-site to control or mitigate the risks during the course of this study:

* The use of standard medical grade materials that have been thoroughly characterized and tested to assure biocompatibility.
* Extensive pre-clinical evaluation including in vitro bench testing and two US FDA IDE studies.
* The well-established transurethral prostatic tissue resection procedure and techniques to be used.
* The ability to quickly and safely abort the study procedure; the physician may elect to discontinue the use of the device at any time in favor of an alternate device/treatment.

E- Ethical oversight:

This study shall be conducted in accordance with the ethical principles that have their origin in the Declaration of Helsinki ("Ethical Principles for Medical Research Involving Human Subjects", 18th World Medical Association General Assembly, Helsinki, Finland, June 1964) and in compliance with the standard ISO 14155:2020 ("Clinical investigation of medical devices for human subjects-Good clinical practice") as well as any regional or national regulations, as appropriate.This study shall not begin until the required approval/favorable opinion from the Ethics Committee or regulatory authority have been obtained, if appropriate. Any additional requirements imposed by the Ethics Committee or regulatory authority shall be followed, if appropriate

F- Data collection and storage: Case report forms (CRFs) will be used to collect all subject data during the study. Data will be stored for 10 years as per institution requirements.

G- Funding: The present study in funded by PROCEPT.

H- Conflict of interest: Although this is an investigator-initiated study, it should be noted that the principal investigator (Dr Naeem Bhojani) is a consultant for PROCEPT.

ELIGIBILITY:
Inclusion Criteria:

* a) Patient has diagnosis of LUTS due to BPH
* b) Patient is mentally capable and willing to sign a study-specific informed consent form
* c) Patient is able and willing to follow study instructions and likely to attend and complete all required study visits

Exclusion Criteria:

* a) Patient is unable to stop anticoagulants, antiplatelet agents, or non-steroidal anti- inflammatory agents (NSAIDs, including aspirin greater or equal to 100mg) prior to treatment per standard of care
* b) Contraindications for general and spinal anesthesia
* c) Patient is unwilling to accept a blood transfusion if required

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
The change of the International Prostate Symptom Score (IPSS) from baseline to 3 months | 3 months
  The International Prostate Symptom Score (IPSS) change from baseline to 3 months will be compared to an objective performance criterion (OPC) based upon published TURP results of 16 points. The IPSS is made up of 7 questions related to voiding symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.
Rate of Unanticipated Serious Adverse Effect (USADE) | Immediately after the surgery
  Unanticipated Serious Adverse Effect (USADE) rate observed up to the 3 months follow-up visit.

SECONDARY OUTCOMES:
Identification of the anatomical landmarks | Immediately after the surgery
  The ability to provide adequate imaging for completing the surgical procedure as assessed by surgeons during the aquablation procedure

OTHER OUTCOMES:
Percentage of study subjects who were discharged on the day of surgery | Immediately after the surgery
  Percentage of study subjects who were discharged on the day of surgery (day case) in subjects ≤ 80 years old with a prostate size ≤150cc , >150cc, and subjects >80 years old with any prostate size
Post-op catheterization duration | 3 months
  Post-op catheterization duration will be calculated
Rate of readmissions within 1 week of discharge | 1 week
  Readmission within 1 week of discharge
Change in uroflow measurements from baseline to 3 month follow up visit | 3 months
  Change in uroflow measurements from baseline to 3 month follow up visit
Operation time | During surgery
  Operation time (TRUS in to catheter in)

CONTACTS AND LOCATIONS:
Overall Officials: Naeem Bhojani, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hunter DJ, McKee CM, Black NA, Sanderson CF. Urinary symptoms: prevalence and severity in British men aged 55 and over. J Epidemiol Community Health. 1994 Dec;48(6):569-75. doi: 10.1136/jech.48.6.569. PMID 7830011
- [Background] Trueman P, Hood SC, Nayak US, Mrazek MF. Prevalence of lower urinary tract symptoms and self-reported diagnosed 'benign prostatic hyperplasia', and their effect on quality of life in a community-based survey of men in the UK. BJU Int. 1999 Mar;83(4):410-5. doi: 10.1046/j.1464-410x.1999.00966.x. PMID 10210562
- [Background] Roehrborn CG, Barkin J, Gange SN, Shore ND, Giddens JL, Bolton DM, Cowan BE, Cantwell AL, McVary KT, Te AE, Gholami SS, Moseley WG, Chin PT, Dowling WT, Freedman SJ, Incze PF, Coffield KS, Herron S, Rashid P, Rukstalis DB. Five year results of the prospective randomized controlled prostatic urethral L.I.F.T. study. Can J Urol. 2017 Jun;24(3):8802-8813. PMID 28646935
- [Background] Gratzke C, Barber N, Speakman MJ, Berges R, Wetterauer U, Greene D, Sievert KD, Chapple CR, Patterson JM, Fahrenkrug L, Schoenthaler M, Sonksen J. Prostatic urethral lift vs transurethral resection of the prostate: 2-year results of the BPH6 prospective, multicentre, randomized study. BJU Int. 2017 May;119(5):767-775. doi: 10.1111/bju.13714. Epub 2016 Dec 21. PMID 27862831
- [Background] Faber K, de Abreu AL, Ramos P, Aljuri N, Mantri S, Gill I, Ukimura O, Desai M. Image-guided robot-assisted prostate ablation using water jet-hydrodissection: initial study of a novel technology for benign prostatic hyperplasia. J Endourol. 2015 Jan;29(1):63-9. doi: 10.1089/end.2014.0304. PMID 25000418
- [Background] Gilling P, Reuther R, Kahokehr A, Fraundorfer M. Aquablation - image-guided robot-assisted waterjet ablation of the prostate: initial clinical experience. BJU Int. 2016 Jun;117(6):923-9. doi: 10.1111/bju.13358. Epub 2015 Nov 19. PMID 26477826
- [Background] Bach T, Giannakis I, Bachmann A, Fiori C, Gomez-Sancha F, Herrmann TRW, Netsch C, Rieken M, Scoffone CM, Tunc L, Rassweiler JJ, Liatsikos E. Aquablation of the prostate: single-center results of a non-selected, consecutive patient cohort. World J Urol. 2019 Jul;37(7):1369-1375. doi: 10.1007/s00345-018-2509-y. Epub 2018 Oct 4. PMID 30288598
- [Background] Gilling P, Anderson P, Tan A. Aquablation of the Prostate for Symptomatic Benign Prostatic Hyperplasia: 1-Year Results. J Urol. 2017 Jun;197(6):1565-1572. doi: 10.1016/j.juro.2017.01.056. Epub 2017 Jan 20. PMID 28111300
- [Background] Misrai V, Rijo E, Zorn KC, Barry-Delongchamps N, Descazeaud A. Waterjet Ablation Therapy for Treating Benign Prostatic Obstruction in Patients with Small- to Medium-size Glands: 12-month Results of the First French Aquablation Clinical Registry. Eur Urol. 2019 Nov;76(5):667-675. doi: 10.1016/j.eururo.2019.06.024. Epub 2019 Jul 5. PMID 31281024
- [Background] Desai M, Bidair M, Zorn KC, Trainer A, Arther A, Kramolowsky E, Doumanian L, Elterman D, Kaufman RP Jr, Lingeman J, Krambeck A, Eure G, Badlani G, Plante M, Uchio E, Gin G, Goldenberg L, Paterson R, So A, Humphreys M, Roehrborn C, Kaplan S, Motola J, Bhojani N. Aquablation for benign prostatic hyperplasia in large prostates (80-150 mL): 6-month results from the WATER II trial. BJU Int. 2019 Aug;124(2):321-328. doi: 10.1111/bju.14703. Epub 2019 Mar 29. PMID 30734990
- [Background] Gilling P, Barber N, Bidair M, Anderson P, Sutton M, Aho T, Kramolowsky E, Thomas A, Cowan B, Kaufman RP Jr, Trainer A, Arther A, Badlani G, Plante M, Desai M, Doumanian L, Te AE, DeGuenther M, Roehrborn C. WATER: A Double-Blind, Randomized, Controlled Trial of Aquablation(R) vs Transurethral Resection of the Prostate in Benign Prostatic Hyperplasia. J Urol. 2018 May;199(5):1252-1261. doi: 10.1016/j.juro.2017.12.065. Epub 2018 Jan 31. PMID 29360529
- [Background] Plante M, Gilling P, Barber N, Bidair M, Anderson P, Sutton M, Aho T, Kramolowsky E, Thomas A, Cowan B, Kaufman RP Jr, Trainer A, Arther A, Badlani G, Desai M, Doumanian L, Te AE, DeGuenther M, Roehrborn C. Symptom relief and anejaculation after aquablation or transurethral resection of the prostate: subgroup analysis from a blinded randomized trial. BJU Int. 2019 Apr;123(4):651-660. doi: 10.1111/bju.14426. Epub 2018 Jul 26. PMID 29862630
- [Background] Sorokin I, Sundaram V, Singla N, Walker J, Margulis V, Roehrborn C, Gahan JC. Robot-Assisted Versus Open Simple Prostatectomy for Benign Prostatic Hyperplasia in Large Glands: A Propensity Score-Matched Comparison of Perioperative and Short-Term Outcomes. J Endourol. 2017 Nov;31(11):1164-1169. doi: 10.1089/end.2017.0489. Epub 2017 Sep 26. PMID 28854815
- [Background] Monn MF, El Tayeb M, Bhojani N, Mellon MJ, Sloan JC, Boris RS, Lingeman JE. Predictors of Enucleation and Morcellation Time During Holmium Laser Enucleation of the Prostate. Urology. 2015 Aug;86(2):338-42. doi: 10.1016/j.urology.2015.04.028. Epub 2015 Jul 15. PMID 26189134
- [Result] TY - JOUR AU - Desai, Mihir AU - Bidair, Mo AU - Bhojani, Naeem AU - Trainer, Andrew AU - Arther, Andrew AU - Kramolowsky, Eugene AU - Doumanian, Leo AU - Elterman, Dean AU - Jr, Ronald AU - Lingeman, James AU - Krambeck, Amy AU - Eure, Gregg AU - Badlani, Gopal AU - Plante, Mark AU - Uchio, Edward AU - Gin, Greg AU - Goldenberg, Larry AU - Paterson, Ryan AU - So, Alan AU - Zorn, Kevin PY - 2018/04/01 SP - T1 - Aquablation Procedural Outcomes for BPH in Large Prostates (80-150cc): Initial Experience VL - 123 DO - 10.1111/bju.14360 JO - BJU International ER -